CLINICAL TRIAL: NCT04148859
Title: Feto-Fetal Transfusion Syndrome in Multiple Pregnancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-220
Record Dates: First submitted 2019-10-20; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Pregnant With Complication
Keywords: TTTS; controlled amnioreduction; amniotic pressure
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: We will recruit 11 women who have to undergo amnioreduction due to TTTS. The amniotic fluid is drained via needle, which is stubbed in the abdomen wall, connected to a tube into a plastic bag. The amniotic fluid pressure will be measured by a water manometer. A T-shape connector will be connected to the tube on one side, and to a short tube on the other side. The height of the fluid within the short tube will indicate the pressure. All the fluid will be drained to the plastic bag. The pressure and the blood flow of the fetuses will be measured during the procedure, depends on the drainage rate. We will include cases of multiple pregnancies with TTTS who must undergo amnioreduction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | US Export: No

ARMS (1):
- pregnant women (Experimental): women who have to undergo amnioreduction due to TTTS
  Interventions: Procedure: amnioreduction

INTERVENTIONS:
Procedure: amnioreduction — The amniotic fluid is drained via needle, which is stubbed in the abdomen wall, connected to a tube into a plastic bag. The amniotic fluid pressure will be measured by a water manometer. A T-shape connector will be connected to the tube on one side, and to a short tube on the other side. The height of the fluid within the short tube will indicate the pressure. All the fluid will be drained to the plastic bag. The pressure and the blood flow of the fetuses will be measured during the procedure, depends on the drainage rate.

SUMMARY:
Objectives: Twin-to-twin transfusion syndrome (TTTS) generates high risk for one of the twins, may lead to preterm delivery and is also associated with neurodevelopmental deficits. The aim of this study was to explore a controlled amnioreduction (AR) procedure in which the amniotic pressure is simultaneously measured with the removed volume of amniotic pressure.

Methods: Eleven patients with severe TTTS at stages II and III of Quintero classification were enrolled to the study. The amniotic pressure was measured along with the removed volume of the amniotic pressure between 17-34 weeks of gestation. The umbilical artery S/D ratio for each twin was measured at the beginning and after every 500cc of removed amniotic fluid. Long-term neurodevelopmental outcome of infants with TTTS was evaluated from a questionnaire for assessing the overall health of the surviving twins.

DETAILED DESCRIPTION:
The placentation of monozygotic twins depends on the stage at which duplication occurs. A monochorionic diamniotic placenta type occurs when the blastocyst splits between days 3 8 after fertilization when the trophoblast but not the amniotic cavity has differentiated. The blood vessels of the twins of such a placenta form superficial or deep anastomoses (Denbow et al., 2000). The anastomoses may communicate between an artery of one twin to an artery of the other one (A-A), vein to vein (V-V) or artery to vein (A-V). The superficial anastomoses are the ones between fairly large vessels on the chorionic plate, where the majority of them are A A. These anastomoses are bidirectional, and allow rapid flow between the twins, depending on pressure gradient. The A-V anastomoses are usually deep and occur in a shared cotyledon where the connection is via the capillary system. These anastomoses are unidirectional and result in an asymmetric flow from one twin to another (Fox, 1997; Bajoria, 1998; Taylor et al, 1999; De Paepe et al, 2002).

Monochorionic diamniotic placentas may be diagnosed by ultrasonography (US) at 8 10 weeks of gestation in the presence of a single placenta, similar genitalia, an intrafetal septum <2 mm thick, and the absence of a twin peak sign (Bajoria, 1998). Twin-twin transfusion syndrome (TTTS) is a major complication of a monochorionic placenta which occurs in 10% 15% of monochorionic multiple pregnancies (Sebire et al, 1997) due to blood transfusion from one twin (the donor) to the other (the recipient) (Bajoria et al, 1995; Talbert et al, 1996). The donor twin becomes anemic and the amount of its amniotic fluid decreases, while the recipient becomes polycythemic, causing polyhydramnios. The cause for the development of TTTS accounts for the types of anastomoses. Mild TTTS has a single deep A V anastomosis along with superficial A-A and V-V anastomoses, whereas severe TTTS lacks the superficial anastomoses (Bajoria, 1998; Denbow et al, 1998; Bermudez et al, 2002). It was postulated that a single, deep A-V anastomosis causes asymmetric blood flow from one twin to the other (3)(Bajoria, 1998). The effect of an asymmetric blood flow is minimized when superficial anastomoses are present together with an A-V anastomosis (Denbow et al, 2000). Superficial anastomoses are clearly observed on the chorionic plate. Deep anastomoses, i.e., the A-V type, represent a shared cotyledon in which the arterial supply is derived from one twin and the venous drainage is to the other (Denbow et al., 1998). Thus, A-V anastomoses may be suspected by an unpaired artery of one twin and an unpaired vein of the other twin being dipped closely into the placenta at a distance <1 cm (De Paepe et al., 2002).

Monochorionic twins have an approximately 25% rate of perinatal morbidity and mortality, which is much higher than singleton and dichorionic twins (Kaufman et al, 1998; De Catte et al., 2002; Chow et al., 2001). No single therapy is associated with a uniformly improved outcome for the involved twins and success is primarily related to gestational age and severity at diagnosis. Treatment options for severe cases include serial amniocenteses, septostomy, laser occlusion of placental vessels, digitalization, ligation of the umbilical cord and selective feticide. These modalities are associated with significant risks of complications, and variable results of fetal morbidity and mortality. Therefore, they should be considered when risks of withholding treatment clearly outweigh those associated with intervention (Ropacka et al, 2002).

The serial amnioreduction is currently the most widely used therapy because it is simple and requires commonly available skilled and equipment. The excess amniotic fluid volume which can vary from 0.5 to few liters are removed, reducing the excess amniotic fluid and pressure, and potentially preventing or delaying rupture of the membranes or preterm labor. Amnioreduction carries a related risk of delivery of 4% per procedure (Van Gemert et al, 2001).

Obliteration of placental anastomoses is the obvious causal therapy of TTTS, because placental anastomoses cause oligo-polyhydramnios sequence of TTTS. The fetoscopic laser coagulates placental vascular anastomoses along the inter-twin septum. However, few anastomoses may be located at the donor side or hidden by the stuck twin and thus, coagulation is limited. TTTS can worsen if compensating vessels (bidirectional) are coagulated instead of significant AV. The risk of procedure-related spontaneous abortion is greater after laser therapy than single amnioreduction. The advantage of amnioreduction changes after three procedures (Van Gemert et al, 2001).

TTTS is not completely understood and is controversial which hampers development of acceptable diagnostic and rational treatment strategies. In this research we would like to investigate the mechanism which improves both twins blood flow after amnioreduction. Such knowledge may improve future management of TTTS. We will recruit 11 women who have to undergo amnioreduction due to TTTS. The amniotic fluid is drained via needle, which is stubbed in the abdomen wall, connected to a tube into a plastic bag. The amniotic fluid pressure will be measured by a water manometer. AT-shape connector will be connected to the tube on one side, and to a short tube on the other side. The height of the fluid within the short tube will indicate the pressure. All the fluid will be drained to the plastic bag. The pressure and the blood flow of the fetuses will be measured during the procedure, depends on the drainage rate. We will include cases of multiple pregnancies with TTTS who must undergo amnioreduction. Pregnancies with malformations or genetic pathologies will be excluded. In addition, we also will explore the long-term neurodevelopmental outcome of children born following a pregnancy complicated by TTTS whose mothers underwent the controlled AR.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancies with TTTS

Exclusion Criteria:

* Pregnancies with malformations or genetic pathologies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 11 (Estimated)
Dates: Start 2004-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The amniotic pressure | The duration of measurements will be about 80 minutes per procedure.
  The amniotic fluid pressure will be measured at the beginning and after every 500cc of removed amniotic fluid by a water manometer. The pattern of the decreasing amniotic pressure during removal of the excess volume of fluid will be depicted.

SECONDARY OUTCOMES:
The removed amniotic volume | The duration of measurements will be about 80 minutes per procedure.
  The removed volume of fluid will be recorded every 500 ml using a sterile bag.
The umbilical artery S/D ratio | The duration of measurements will be about 80 minutes per procedure.
  The umbilical artery S/D ratio for each twin will be measured with a Doppler ultrasound machine at the beginning and after every 500cc of removed amniotic fluid. The graph of the umbilical artery S/D ratio vesus weeks of gestation will be plotted.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel J Jaffa, MD, Principal Investigator — Ultrasound Unit in Obstetrics and Gynecology, Lis Maternity Hospital
Locations (1):
- Zoya Gordon, Tel Aviv, Israel